CLINICAL TRIAL: NCT00736437
Title: Efficacy of Acyclovir in Combination With a Glucocorticosteroid on UV-Induced Herpes Labialis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Borje Darpo, MD, PhD, Medivir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-609-013
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Herpes Labialis
Keywords: UV-induced; Herpes labialis; time to healing
MeSH Terms: conditions — Herpes Labialis | interventions — ME 609

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ME-609
  Interventions: Drug: ME-609
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ME-609 — Cream applied topically 6 times daily over the UVR exposed area
  Arms: 1
Drug: Vehicle — Treatment applied 6 times daily over the UVR exposed area
  Arms: 2

SUMMARY:
The primary objective was to compare the efficacy of ME-609 cream vs placebo cream on the time to healing (loss of hard crust) of delayed classical herpes labialis (HSV) lesions experimentally induced after ultra violet radiation (UVR) exposure.

DETAILED DESCRIPTION:
The primary objective was to compare the efficacy of ME-609 cream vs placebo cream on the time to healing (loss of hard crust) of delayed classical herpes labialis (HSV) lesions experimentally induced after ultra violet radiation (UVR) exposure. Secondary objectives were to compare the time to normal skin, incidence of lesion development (number and type of lesions), maximum lesion size, length of lesion stages, frequency/severity/duration of pain, frequency/severity/duration of tenderness, redness and/or oedema in the UVR exposed area, frequency of virus positive lesions, time to cessation of viral shedding and safety of ME-609 cream vs placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* A history of reactivation of recurrent herpes labialis with overexposure to sunlight in the last 12 months, or 2 or more cold sore lesions in the last 12 months
* Generally healthy as determined by medical history and verbal interview
* Females who were still able to conceive were to have had a negative pregnancy test on enrolment
* Fritzpatrick skin type category of I to IV

Exclusion Criteria:

* Previous inclusion in this study

  * Participation in clinical investigational drug studies in the 4-week period prior to enrolment
  * Participation in any herpes UVR reactivation study within the previous 3 months
  * Previous herpes vaccination at any time
  * Occurrence of herpes labialis (end of episode) within one month prior to enrolment
  * Inflammatory, congenital or iatrogenic underlying immunodeficiency disorders
  * Use of topical steroids in or near the face or on the forearms, systemic steroids (within 30 days from enrolment) or anti-inflammatory drugs (within 10 days from enrolment)
  * Women who were pregnant, lactating or breast feeding
  * Women of child bearing potential not using adequate contraception as judged by the investigator
  * Recent history of alcohol or drug abuse which in the opinion of the investigator could interfere with compliance
  * Significant skin disease such as atopic dermatitis or eczema, that would interfere with the assessment of lesions
  * Allergy or hypersensitivity to steroids, acyclovir, penciclovir and/or other nucleoside analogues
  * Administration of any drug commonly associated with photosensitivity (tetracycline, Retin A) within one week of UVR exposure
  * Any antiviral therapy within 14 days prior to enrolment
  * History of allergy or sensitivity to sunscreen
  * History of herpes keratitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 1999-08; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
time to healing (loss of hard crust) of delayed classical herpes labialis (HSV) lesions experimentally induced after ultra violet radiation (UVR) exposure. | 5 days

SECONDARY OUTCOMES:
time to normal skin, incidence of lesion development, max lesion size, length of lesion stages, pain and tenderness, redness and/or oedema in the UVR exposed area, frequency of virus positive lesions, time to cessation of viral shedding and safety | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Spotswood L Spruance, MD, Principal Investigator — University of Utah